CLINICAL TRIAL: NCT02332551
Title: A Prospective Clinical Trial Using Irreversible Electroporation (IRE) for the Treatment of Unresectable Hepatic Carcinoma Close to the Gallbladder
Brief Title: Percutaneous Irreversible Electroporation to Treat Liver Cancer Close to the Gallbladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JF-20141229
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2019-04

CONDITIONS: Hepatic Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NanoKnife IRE System (Experimental): 90 pulses of 70 microseconds each in duration will be administered per electrode pair
  Interventions: Device: NanoKnife
- Control (No Intervention)

INTERVENTIONS:
Device: NanoKnife — Irreversible electroporation (IRE) is a new, minima-invasive image-guided treatment method for tumors not amenable for surgical resection or thermal ablation, due to vicinity near vital structures such as vessels,bile ducts and the gallbladder .
  Other Names: IRE
  Arms: NanoKnife IRE System

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of irreversible electroporation for unresectable Hepatic carcinoma close to the gallbladder, also Progress Free Survival (PFS) will be recorded.

DETAILED DESCRIPTION:
Hepatic carcinoma is the fifth most common cancer worldwide and a large proportion of patients are unsuitable for tumor resection because of factors such as poor hepatic reserve(cirrhosis), multicentric tumors or near vital structures such as vessels, diaphragmatic dome and gallbladder. Direct ablative treatments include radiofrequency ablation, microwave (MW) ablation and cryotherapy and irreversible electroporation had been used successful as a therapeutic choice for unresectable patients. At the same time，Irreversible electroporation(IRE)，which was applied with a novel ablation technology, can induce tissue necrosis by utilizing short pulses of high-voltage electrical energy. The technique also had many advantages, including Short ablation time, preservation of vital structures within IRE-ablated zone, avoidance of heat/cold-sink effect, complete ablation with well-demarcated margin and real-time monitoring of IRE ablation.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic carcinoma diagnosed by positive biopsy or non-invasive criteria,
* Tumor from gallbladder is <0.5 cm
* not suitable for surgical resection or transplantation,
* have at least one, but less than or equal to 3 tumors,
* of the tumour(s) identified, each tumor must be ≤ 7 cm in diameter,
* Child-Pugh class A,B
* Eastern Cooperative Oncology Group (ECOG) score of 0-1,
* American Society of Anaesthesiologists (ASA) score ≤ 3,
* a prothrombin time ratio > 50%,
* platelet count > 80x109/L,
* ability of patient to stop anticoagulant and anti-platelet therapy for seven days prior to and seven days post NanoKnife procedure,
* are able to comprehend and willing to sign the written informed consent form (ICF),
* have a life expectancy of at least 3 months.

Exclusion Criteria:

* eligible for surgical treatment or transplantation for HCC,
* Hepatic carcinoma developed on an already transplanted liver,
* cardiac insufficiency, ongoing coronary artery disease or arrhythmia,
* any active implanted device (eg Pacemaker),
* women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
* have received treatment with an investigational agent/ procedure within 30 days prior to treatment with the NanoKnife™ LEDC System, are in the opinion of the Investigator unable to comply with the visit schedule and protocol evaluations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy as measured by modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria by Computed Tomography (CT) or Magnetic Resonance (MR) imaging. | 30 days (+/- 3 days) post treatment

SECONDARY OUTCOMES:
Safety using Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 criteria. | Immediately post treatment to 2 years post treatment

OTHER OUTCOMES:
Progress free survival(PFS) | 24months

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi l Niu, PHD, Study Chair — FUDA Cancer Hospital
Locations (1):
- 中国, Guangzhou, Guangdong, China